Statistical Analysis Plan for Protocol

Status: Approved, Version: 2.0

Approved Date: 13 Jan 2021

CLL949-E003 / NCT04702984

This version of the Statistical Analysis Plan is based on Version 1.0 of the study protocol.

C-CLN-0004795 Approved Date: 13 Jan 2021

#### **Executive Summary:**

Key Objective:

The primary objective of this study is to evaluate the clinical performance of an investigational frequent replacement daily wear silicone hydrogel (SiHy) sphere contact lens, over 7 days of daily wear.


Decision Criteria for Study Success:

Decision criteria for study success are not applicable for this study.

### **Table of Contents**

| Sta | itistical Ai | nalysis Plan for Protocol CLL949-E003 | 1 |
|---|---|---|---|
| Tal | ole of Cor | itents | 3 |
| Lis | st of Table | S | |
| 1 | | ojectives and Design | |
| | 1.1 | Study Objectives | |
| | 1.1 | Study Objectives | |
| | 1.3 | Randomization | |
| | 1.3 | Masking | |
| | 1.4 | Widsking | |
| 2 | Analysis | Sets | 6 |
| | 2.1 | Safety Analysis Set | |
| 3 | | Characteristics and Study Conduct Summaries | |
| 4 | Effectiveness Analysis Strategy | | |
| | 4.1 | Effectiveness Endpoints | |
| | 4.2 | Effectiveness Hypotheses | |
| | 4.3 | Statistical Methods for Effectiveness Analyses | |
| | 1.5 | 4.3.1 Primary Effectiveness Analyses | |
| 5 | Safety A | nalysis Strategy | 9 |
| | 5.1 | Safety Endpoints | 9 |
| | 5.2 | Safety Hypotheses | 10 |
| | 5.3 | Statistical Methods for Safety Analyses | 10 |
| | | 5.3.1 Adverse Events | 10 |
| | | 5.3.2 Biomicroscopy Findings/Slit Lamp Examination | |
| _ | | 5.3.3 Device Deficiencies | 11 |

| Document ID:<br>V-CLN-0004795 | | Status: Approved, Version: 2.0<br>Approved Date: 13 Jan 2021 | Page 4 of 15 |
|---|---|---|---|
| 8 Referen | ces | | 11 |
| 9 Revision | ı History | | 12 |
| 9.1 | Amendment 1 (Version | n 2.0) | 12 |
| 10 Append | ix | | 13 |
| T 11 1 1 | g, 1 D | List of Tables | - |
| Table 1-1 | Study Description Su | mmary | 5 |

Table 10-1

Status: Approved, Version: 2.0 Approved Date: 13 Jan 2021

# 1 Study Objectives and Design

# 1.1 Study Objectives

The primary objective of this study is to evaluate the clinical performance of an investigational frequent replacement daily wear SiHy sphere contact lens, over 7 days of daily wear.

# 1.2 Study Description

Key components of the study are summarized in Table 1-1.

Table 1-1 Study Description Summary

| Study Design | Prospective, single group, bilateral, open-label |
|---|---|
| Study Population | Volunteer subjects aged 18 or over who are habitual spherical |
| | daily wear soft frequent replacement contact lens wearers, have |
| | at least 3 months of contact lens wearing experience, and who |
| | wear their habitual lenses at least 5 days per week for at least 8 |
| | hours per day. |
| | Target to complete: 30 |
| | Planned to enroll: ~ 48 |
| Number of Sites | ~3 |
| | US |
| Test Product | LID021201 |
| Control Product | N/A |
| Duration of Treatment | Test Product: ~ 7 days |
| Visits | Visit 1 – Screening/Baseline/Order Spectacles |
| | Visit 2 — Dispense Study Lens |
| | Visit 3 Week 1 Follow-up/Exit |

1.3 Randomization

Randomization is not applicable for this study.

#### 1.4 Masking

This is a single group, open-label study.

### 2 Analysis Sets

### 2.1 Safety Analysis Set

Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis. As such, the safety analysis set will include all subjects/eyes exposed to any study lenses evaluated in this study, except for the lenses used with the purpose of over-spectacle determination.


Approved Date: 13 Jan 2021

For treatment-emergent safety analyses, subjects/eyes will be categorized under the actual study lenses exposed.

Adverse events occurring from the time of informed consent but prior to first exposure to study lenses will be summarized in subject listings.

# **3** Subject Characteristics and Study Conduct Summaries

The following tables will be presented:

- Subject Disposition
- Analysis Set
- Subject Accounting
- Demographics Characteristics
- Baseline Characteristics [eg, lens brand, lens care brand]



Approved Date: 13 Jan 2021 **Effectiveness Analysis Strategy** 4 This study defines one primary endpoint Safety Analysis Set will be used for all effectiveness analyses. All data obtained in evaluable subjects/eyes will be included in the analysis. No imputation for missing values will be carried out. 4.1 **Effectiveness Endpoints Primary Endpoint** The primary endpoint is front surface wettability, collected on a 5-point scale, for each eye.




# **4.2** Effectiveness Hypotheses

#### **Primary Effectiveness**

No inferences are to be made on the primary effectiveness endpoint; therefore, no hypotheses are formulated.




Page 9 of 15

# 4.3 Statistical Methods for Effectiveness Analyses

### 4.3.1 Primary Effectiveness Analyses

Descriptive statistics will be presented, to include frequencies and percentages in each grade as well as for the combined category of Grade 0 and Grade 1.


Approved Date: 13 Jan 2021



# 5 Safety Analysis Strategy

The focus of the safety analysis will be a comprehensive descriptive assessment of occurrence of adverse events as well as the other listed parameters. Therefore, no inferential testing will be done for the safety analysis.

# 5.1 Safety Endpoints

The safety endpoints are:

- Adverse events (AE)
- Biomicroscopy Findings/Slit Lamp Examinations



• Device deficiencies

### 5.2 Safety Hypotheses

There are no formal safety hypotheses in this study. The focus of the safety analysis will be a comprehensive descriptive assessment of safety endpoints listed in Section 5.1.


Approved Date: 13 Jan 2021

# 5.3 Statistical Methods for Safety Analyses

The analysis set for all safety analyses is defined in Section 2.1.

#### **5.3.1** Adverse Events

The applicable definition of an AE is in the study protocol. All AEs occurring from when a subject signs informed consent to when a subject exits the study will be accounted for in the reporting.

Pre-treatment AEs will be separated from treatment-emergent AEs occurring during the study period. A pre-treatment AE is an event that occurs after signing informed consent but prior to exposure to study lenses. The period for treatment-emergent AE analysis starts from exposure to study lenses until the subject completes or is discontinued from the study.





#### **5.3.3** Device Deficiencies

The following tables and supportive listings will be provided:

- Frequency of Treatment-Emergent Device Deficiencies
- Listing of Treatment-Emergent Device Deficiencies
- Listing of Device Deficiencies Prior To Treatment Exposure



#### **8** References

Not applicable.

Status: Approved, Version: 2.0 Approved Date: 13 Jan 2021

# 9 Revision History

This is Version 2.0 of the Statistical Analysis Plan for this study. This version of the Statistical Analysis Plan is based on Version 1.0 of the study protocol.

### 9.1 Amendment 1 (Version 2.0)

<u>Purpose of Amendment:</u> The purpose of this amendment is detailed below:

• Added sub-bullet in Section 4.1, Exploratory Endpoints

# 10 Appendix

Table 10-1 Schedule of Study Procedures and Assessments


Approved Date: 13 Jan 2021

| Procedure/ Assessment | Visit 1<br>Screening/<br>Baseline/ | Visit 2†<br>Dispense | Visit 3<br>Week 1<br>Follow-up/<br>Exit | Early Exit | USV |
|---|---|---|---|---|---|
| Informed Consent | ✓ | | _ | _ | _ |
| Demographics | ✓ | _ | _ | _ | _ |
| Medical History* | ✓ | <b>√*</b> * | <b>√</b> | <b>√</b> | <b>√</b> |
| Concomitant Medications* | ✓ | <b>√*</b> * | ✓ | ✓ | ✓ |
| Inclusion/Exclusion | ✓ | - | _ | _ | - |
| Habitual lens | | | | | |
| (brand, power* and | ✓ | - | - | - | - |
| lenscare) | | | | | |
| Biomicroscopy | ✓ | <b>√*</b> * | ✓ | <b>✓</b> | <b>√</b> |
| | | | | | _ |
| Record study lens power | ✓ | - | - | - | - |
| Dispense study lenses*∞ | • | ✓ | - | - | - |

| Procedure/ Assessment | Visit 1<br>Screening/<br>Baseline/<br>Order<br>Spectacles | Visit 2†<br>Dispense | Visit 3<br>Week 1<br>Follow-up/<br>Exit | Early Exit | USV |
|---|---|---|---|---|---|
| Lens surface assessments | | | | | |
| (OD, OS): | | | | | |
| Front surface wettability | - | √ | ✓ | ✓ | (✓) |

| Procedure/ Assessment | Visit 1<br>Screening/<br>Baseline/<br>Order<br>Spectacles | Visit 2†<br>Dispense | Visit 3<br>Week 1<br>Follow-up/<br>Exit | Early Exit | USV |
|---|---|---|---|---|---|
| AEsΩ | ✓ | ✓ | ✓ | ✓ | ✓ |
| Device deficiencies | <b>√</b> | <b>√</b> | <b>√</b> | <b>√</b> | ✓ |
| Exit Form | (^) | (√) | <b>√</b> | <b>(√)</b> | (√) |

